CLINICAL TRIAL: NCT06814028
Title: Transcutaneous Auricular Neurostimulation as a Treatment for Women With Heavy Menstrual Bleeding: A Dose-finding Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Biomedical, Inc. (Industry)
Collaborators: Five Liters, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5L-BLD-07
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Heavy Menstrual Bleeding
Keywords: Neurostimulation; Hemostasis; Menstrual cycle; Menstruation; Blood loss; PBAC; Menorrhagia; CMSS; Transcutaneous Auricular Neurostimulation; tAN; Heavy menstrual bleeding
MeSH Terms: conditions — Menorrhagia; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Participants with idiopathic HMB will be enrolled in the study over the course of three consecutive menstrual cycles. First Menstruation will be baseline. The Second Menstruation participants will self-administer 2, 1-hour sessions of active tAN daily beginning Day 1 of menstruation through the final day of menstruation. The Third Menstruation participants will self-administer 1, 2-hour session of active tAN daily beginning Day 1 of menstruation through the final day of menstruation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Heavy Menstrual Bleeding Patients (Experimental): Participants with no known cause of HMB who are not on hormonal therapy. First Menstruation (baseline/no active tAN) followed by Second Menstruation (2 one-hour active tAN sessions daily) followed by Third Menstruation (1 two-hour active tAN session daily).
  Interventions: Device: Volta System

INTERVENTIONS:
Device: Volta System — The Volta System will be using the components of the Sparrow Ascent device: (FDA-cleared K230796) a wearable, battery-operated, neurostimulation system designed to transcutaneously stimulate nerves on and/or around the auricle. During the Second and Third Menstruations, participants will self-administer daily active tAN sessions Volta System Device beginning Day 1 of menstruation through the final day of menstruation.

SUMMARY:
This study is designed as an open label, single-arm, decentralized research study in which patients with idiopathic heavy menstrual bleeding will receive transcutaneous auricular neurostimulation (tAN), which targets the auricular branch of the vagus nerve (ABVN) and the auriculotemporal nerve (ATN). Participants will be enrolled over the course of three menstruations: one baseline menstruation and two menstruations with added daily neurostimulation.

DETAILED DESCRIPTION:
This study is designed as an open label, single arm, cross-over decentralized clinical study in which patients with idiopathic heavy menstrual bleeding will receive transcutaneous auricular neurostimulation (tAN), which targets the auricular branch of the vagus nerve (ABVN) via the mastoid and the auriculotemporal nerve (ATN) anterior to the tragus. Participants will be enrolled into the study over the course of three consecutive menstrual cycles.

During the First Menstruation (baseline), no tAN treatment will be delivered. Participants will estimate blood loss using the Pictorial Bleeding Assessment Chart (PBAC) daily throughout the duration of the menstruation phase of their menstrual cycle. Menstrual symptoms will be assessed using the Cox Menstrual Symptom Scale (CMSS) and a general quality of life assessment will be conducted on the final day of menstruation using the Short-Form 36 (SF-36).

During the Second Menstruation, participants will self-administer two 1-hour active tAN sessions daily (once in the AM, once in the PM), beginning Day 1 of menstruation through the final day of menstruation. Blood loss will be assessed daily using the PBAC throughout the duration of menstruation. Quality of life will be assessed with the CMSS and SF-36 on the final day of menstruation.

During the Third Menstruation, participants will self-administer a single 2-hour active tAN session each day, beginning Day 1 of menstruation through the final day of menstruation. Blood loss will be assessed daily using the PBAC throughout the duration of menstruation. Quality of life will be assessed with the CMSS and SF-36 on the final day of menstruation.

In addition, a device satisfaction survey will be completed at the end of the study. Participants will exit the study after the final day of their third menstruation.

ELIGIBILITY:
Inclusion Criteria:

1. Regularly menstruating female participants between 18-45 years of age
2. History of menorrhagia as assessed by the Menorrhagia Screening Tool
3. Stable/consistent use of current medications and supplements for the past three months, willingness to continue use for duration of study, and not start any new medications or homeopathic remedies
4. Reliable access to an internet-enabled device to complete required questionnaires
5. Willingness to consistently use the same brand of tampons and/or pads throughout duration of the study

Exclusion Criteria:

1. Pregnancy within three months of enrollment
2. Lactating at the time of enrollment
3. Typical length of menstruation greater than 14 days
4. Use of hormone therapy in the past three months
5. Antifibrinolytic use within 30 days of enrollment
6. Known inherited or acquired bleeding disorder
7. Use of anticoagulants (i.e., Aspirin, Warfarin, Coumadin, etc.) including platelet inhibitors for 30 days prior to enrollment
8. Use of the Copper intrauterine device within the past 3 months
9. Known structural cause of heavy menstrual bleeding
10. Use of menstrual cups or menstrual underwear as a method of menstrual blood collection
11. Participant has a history of chronic tobacco use or has ingested nicotine via smoking, vaping, smokeless tobacco, or nicotine patches in the past three months
12. Participant has received a blood transfusion within 30 days prior to study
13. Participant has a history of epileptic seizures
14. Participant has a history of neurologic diseases or traumatic brain injury
15. Participant has presence of devices (e.g., pacemakers, cochlear prostheses, neurostimulators)
16. Participant has abnormal ear anatomy or ear infection present
17. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants are risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Regularly menstruating females.
Enrollment: 40 (Actual)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Blood loss | Daily throughout all three menstruations (up to 3 complete menstrual cycles - estimated 90 days)
  Comparison of mean Pictorial Bleeding Assessment Chart (PBAC) scores during first menstruation (no stimulation) versus second and third menstruations (active stimulation). The PBAC is a widely accepted tool for patients with HMB to account for menstrual blood loss. Menstrual blood loss is estimated through a selection of images of tampons, pads, clots, and flooding events. Patients mark a tally next to the images that best match each of the menstruation products they used that day.
Quality of life | Final day of each menstruation (up to 3 complete menstrual cycles - estimated 90 days)
  Comparison of mean quality of life score measured by the Short Form 36 (SF-36) during first menstruation (no stimulation) versus second and third menstruations (active stimulation). The SF-36 is a 36-item patient-reported questionnaire that assesses general quality of life. This questionnaire includes eight variables: physical functioning, social functioning, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy and vitality, pain, and general perception of health. The SF-36 is scored using a standardized scoring algorithm or by the SF-36 scoring software. The SF-36 scores range from 0 to 100, with higher scores representing better health status.
Duration and severity of dysmenorrhea | Final day of each menstruation (up to 3 complete menstrual cycles - estimated 90 days)
  Comparison of mean Cox Menstrual Symptom Scale (CMSS) scores during first menstruation (no stimulation) versus second and third menstruations (active stimulation). The CMSS measures menstrual distress and dysmenorrhea. The CMSS Severity subscale is an 18-item self-reported scale that measures severity of menstrual symptoms, including pain, nausea, emotions, etc. during menstruation. The CMSS will be used in this trial to measure a participant's dysmenorrhea every day of each menstruation. Each CMSS item is scored from 0-4, with a higher score indicating higher dysmenorrhea severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Five Liters - DECENTRALIZED STUDY, Dallas, Texas, United States